CLINICAL TRIAL: NCT02451137
Title: A Randomized, Open-label, Parallel Group Real World Pragmatic Trial to Assess the Clinical and Health Outcomes of Toujeo Compared to Commercially Available Basal Insulins for Initiation of Therapy in Insulin-naive Patients With Uncontrolled Type 2 Diabetes Mellitus
Brief Title: A "Real World" Trial to Determine Efficacy and Health Outcomes of Toujeo (ACHIEVE CONTROL REAL LIFE STUDY PROGRAM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS14347; U1111-1168-0354 (Other: UTN)
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Toujeo (Experimental): Toujeo® (Insulin glargine, 300 units per millilitre [U/mL]) subcutaneous (SC) injection once daily up to Month 12, with or without available participant support program.
  Interventions: Drug: Insulin glargine, 300 U/ml; Drug: Background Therapy
- Standard of Care (Active Comparator): Lantus® (Insulin glargine, 100 U/mL) SC injection administered once daily; or Levemir® (Insulin detemir) SC injection administered either once or twice daily up to Month 12, with or without available participant support program.
  Interventions: Drug: Insulin glargine, 100 U/ml; Drug: Insulin detemir; Drug: Background Therapy

INTERVENTIONS:
Drug: Insulin glargine, 300 U/ml — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: Toujeo
  Arms: Toujeo
Drug: Insulin glargine, 100 U/ml — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: Lantus
  Arms: Standard of Care
Drug: Insulin detemir — Pharmaceutical form: solution
  Route of administration: subcutaneous
  Other Names: Levemir
  Arms: Standard of Care
Drug: Background Therapy — Anti-diabetic drugs at investigator discretion and consistent with local labeling guidelines for use with insulin.

SUMMARY:
Primary Objective:

Demonstrate clinical benefit of Toujeo in achieving individualized Healthcare Effectiveness Data and Information Set (HEDIS) glycated hemoglobin (HbA1c) targets (<8% if age >=65 years or with defined comorbidities or otherwise <7%) at 6 months without documented symptomatic (Blood Glucose <=70 mg/deciliter [mg/dL]) and/or severe hypoglycemia at any time of day from baseline to 6 months in uncontrolled insulin naive participants with type 2 diabetes initiating basal insulin therapy in a real world setting.

Secondary Objectives:

Compare Toujeo to other commercially available basal insulins at 6 months after initiating insulin therapy in a real world setting in terms of:

* Participant persistence with assigned basal insulin therapy.
* Risk of hypoglycemia including the incidence and rate of documented symptomatic and severe hypoglycemia.
* Changes in HbA1c, fasting plasma glucose, body weight
* Differences in participant and provider- reported outcomes (including Diabetes Treatment Satisfaction Questionnaire Status and Change Versions (DTSQs) and (DTSQc), Hypoglycemia Patient Questionnaire, and participant and provider reported Global Effectiveness Scale (GES).
* Healthcare resource utilization including hospitalizations and emergency department or other provider visits and healthcare costs.

DETAILED DESCRIPTION:
The total study duration per patient will be up to 53 weeks, consisting of a 1-week screening period at the site, a 26-week treatment period, and a 26-week extension period.

ELIGIBILITY:
Inclusion criteria :

* Participants with Type 2 Diabetes Mellitus (T2DM), as defined by the American Diabetes Association/World Health Organization, diagnosed for at least 1 year at the time of the screening visit, insufficiently controlled after at least 1 year of treatment with 2 or more of the following: oral agents (metformin, sulfonylureas, thiazolidinediones, dipeptidyl peptidase-4 (DPP4) inhibitors, or sodium-glucose cotransporter 2 (SGLT2) inhibitors) or glucagon-like peptide-1 (GLP-1) receptor agonists approved for daily use with insulin (Victoza, Byetta, Adlyxin).
* Adult patients who have signed an Informed Consent Form and Health Insurance Portability and Accountability Act (HIPAA) Authorization Form.

Exclusion criteria:

* HbA1c <8.0% or >11.0%.
* Males or females <18 years of age.
* Type 1 diabetes mellitus.
* Any clinically significant abnormality identified on physical examination, laboratory tests, or vital signs at the time of screening, or any major systemic disease resulting in short life expectancy that in the opinion of the Investigator would restrict or limit the participant's successful participation for the duration of the study.
* Use of any product containing insulin (Lantus, Levemir, Humulin, Novolin, Humalog, Novolog, Apidra, or Afrezza) since the time of diagnosis with T2DM other than temporary use during pregnancy or hospitalization, or short-term use during acute event.
* Use of oral hypoglycemic agents other than those noted in the inclusion criteria, GLP-1 receptor agonists for weekly use, or any investigational agent (drug, biologic, or device) within 3 months prior to the time of screening.
* All contraindications to commercially available insulin therapy or warnings/precautions of use as displayed in the respective national product labeling for these products.
* Pregnancy or lactation.
* Women of childbearing potential with no effective contraceptive method.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3304 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (427):
- United States (407):
  - Investigational Site Number 840731, Birmingham, Alabama
  - Investigational Site Number 840305, Birmingham, Alabama
  - Investigational Site Number 840811, Birmingham, Alabama
  - Investigational Site Number 840218, Gulf Shores, Alabama
  - Investigational Site Number 840739, Guntersville, Alabama
  - Investigational Site Number 840367, Huntsville, Alabama
  - Investigational Site Number 840130, Montgomery, Alabama
  - Investigational Site Number 840729, Montgomery, Alabama
  - Investigational Site Number 840281, Saraland, Alabama
  - Investigational Site Number 840613, Sheffield, Alabama
  - Investigational Site Number 840634, Sheffield, Alabama
  - Investigational Site Number 840654, Sheffield, Alabama
  - Investigational Site Number 840173, Phoenix, Arizona
  - Investigational Site Number 840555, Phoenix, Arizona
  - Investigational Site Number 840805, Sun City, Arizona
  - Investigational Site Number 840725, Conway, Arkansas
  - Investigational Site Number 840790, Jonesboro, Arkansas
  - Investigational Site Number 840699, Little Rock, Arkansas
  - Investigational Site Number 840528, Little Rock, Arkansas
  - Investigational Site Number 840079, Searcy, Arkansas
  - Investigational Site Number 840337, Bakersfield, California
  - Investigational Site Number 840089, El Cajon, California
  - Investigational Site Number 840024, Escondido, California
  - Investigational Site Number 840020, Fresno, California
  - Investigational Site Number 840470, Imperial, California
  - Investigational Site Number 840155, Inglewood, California
  - Investigational Site Number 840161, Inglewood, California
  - Investigational Site Number 840194, Laguna Hills, California
  - Investigational Site Number 840710, Laguna Hills, California
  - Investigational Site Number 840204, Lancaster, California
  - Investigational Site Number 840371, Los Angeles, California
  - Investigational Site Number 840310, Los Angeles, California
  - Investigational Site Number 840504, Los Angeles, California
  - Investigational Site Number 840340, Los Angeles, California
  - Investigational Site Number 840309, Los Gatos, California
  - Investigational Site Number 840256, North Hollywood, California
  - Investigational Site Number 840015, Northridge, California
  - Investigational Site Number 840056, Norwalk, California
  - Investigational Site Number 840090, Orange, California
  - Investigational Site Number 840078, Palm Springs, California
  - Investigational Site Number 840791, Palmdale, California
  - Investigational Site Number 840216, Paramount, California
  - Investigational Site Number 840413, Pomona, California
  - Investigational Site Number 840244, Port Hueneme, California
  - Investigational Site Number 840162, San Diego, California
  - Investigational Site Number 840028, San Diego, California
  - Investigational Site Number 840383, San Dimas, California
  - Investigational Site Number 840627, San Jose, California
  - Investigational Site Number 840120, San Ramon, California
  - Investigational Site Number 840156, Santa Ana, California
  - Investigational Site Number 840266, Sherman Oaks, California
  - Investigational Site Number 840091, Sylmar, California
  - Investigational Site Number 840208, Thousand Oaks, California
  - Investigational Site Number 840115, Torrance, California
  - Investigational Site Number 840792, Torrance, California
  - Investigational Site Number 840612, Tulare, California
  - Investigational Site Number 840467, Upland, California
  - Investigational Site Number 840185, Vista, California
  - Investigational Site Number 840472, Whittier, California
  - Investigational Site Number 840411, Aurora, Colorado
  - Investigational Site Number 840596, Denver, Colorado
  - Investigational Site Number 840170, Denver, Colorado
  - Investigational Site Number 840188, Englewood, Colorado
  - Investigational Site Number 840329, Littleton, Colorado
  - Investigational Site Number 840728, Littleton, Colorado
  - Investigational Site Number 840687, Northglenn, Colorado
  - Investigational Site Number 840643, Aventura, Florida
  - Investigational Site Number 840652, Boca Raton, Florida
  - Investigational Site Number 840449, Bradenton, Florida
  - Investigational Site Number 840081, Cooper City, Florida
  - Investigational Site Number 840027, Coral Gables, Florida
  - Investigational Site Number 840446, Coral Gables, Florida
  - Investigational Site Number 840407, Cutler Bay, Florida
  - Investigational Site Number 840083, Doral, Florida
  - Investigational Site Number 840141, Fleming Island, Florida
  - Investigational Site Number 840035, Fort Lauderdale, Florida
  - Investigational Site Number 840068, Fort Lauderdale, Florida
  - Investigational Site Number 840145, Hialeah, Florida
  - Investigational Site Number 840142, Jacksonville, Florida
  - Investigational Site Number 840352, Jacksonville, Florida
  - Investigational Site Number 840021, Jupiter, Florida
  - Investigational Site Number 840639, Kissimmee, Florida
  - Investigational Site Number 840640, Kissimmee, Florida
  - Investigational Site Number 840777, Lake Clarke Shores, Florida
  - Investigational Site Number 840362, Margate, Florida
  - Investigational Site Number 840002, Miami, Florida
  - Investigational Site Number 840012, Miami, Florida
  - Investigational Site Number 840698, Miami, Florida
  - Investigational Site Number 840102, Miami, Florida
  - Investigational Site Number 840209, Miami, Florida
  - Investigational Site Number 840014, Miami, Florida
  - Investigational Site Number 840128, Miami, Florida
  - Investigational Site Number 840143, Miami, Florida
  - Investigational Site Number 840349, Miami, Florida
  - Investigational Site Number 840758, Miami, Florida
  - Investigational Site Number 840690, Miami, Florida
  - Investigational Site Number 840415, Miami, Florida
  - Investigational Site Number 840197, Miami, Florida
  - Investigational Site Number 840414, Miami, Florida
  - Investigational Site Number 840221, Miami Lakes, Florida
  - Investigational Site Number 840303, Miami Lakes, Florida
  - Investigational Site Number 840508, Ocala, Florida
  - Investigational Site Number 840092, Ocoee, Florida
  - Investigational Site Number 840118, Palm Harbor, Florida
  - Investigational Site Number 840080, Panama City, Florida
  - Investigational Site Number 840372, Plantation, Florida
  - Investigational Site Number 840199, Port Charlotte, Florida
  - Investigational Site Number 840538, Winter Haven, Florida
  - Investigational Site Number 840261, Atlanta, Georgia
  - Investigational Site Number 840232, Atlanta, Georgia
  - Investigational Site Number 840129, Blue Ridge, Georgia
  - Investigational Site Number 840820, Columbus, Georgia
  - Investigational Site Number 840767, Decatur, Georgia
  - Investigational Site Number 840812, Decatur, Georgia
  - Investigational Site Number 840700, Dunwoody, Georgia
  - Investigational Site Number 840648, East Point, Georgia
  - Investigational Site Number 840110, Lawrenceville, Georgia
  - Investigational Site Number 840444, Macon, Georgia
  - Investigational Site Number 840003, Marietta, Georgia
  - Investigational Site Number 840632, Sandersville, Georgia
  - Investigational Site Number 840616, Savannah, Georgia
  - Investigational Site Number 840591, Savannah, Georgia
  - Investigational Site Number 840727, Smyrna, Georgia
  - Investigational Site Number 840520, Snellville, Georgia
  - Investigational Site Number 840163, Statesboro, Georgia
  - Investigational Site Number 840297, Stockbridge, Georgia
  - Investigational Site Number 840715, Thomson, Georgia
  - Investigational Site Number 840400, Blackfoot, Idaho
  - Investigational Site Number 840764, Boise, Idaho
  - Investigational Site Number 840005, Chicago, Illinois
  - Investigational Site Number 840399, Chicago, Illinois
  - Investigational Site Number 840301, Elgin, Illinois
  - Investigational Site Number 840402, Joliet, Illinois
  - Investigational Site Number 840226, Morton, Illinois
  - Investigational Site Number 840318, Peoria, Illinois
  - Investigational Site Number 840125, Avon, Indiana
  - Investigational Site Number 840344, Brownsburg, Indiana
  - Investigational Site Number 840007, Evansville, Indiana
  - Investigational Site Number 840164, Evansville, Indiana
  - Investigational Site Number 840324, Evansville, Indiana
  - Investigational Site Number 840022, Franklin, Indiana
  - Investigational Site Number 840536, Greenfield, Indiana
  - Investigational Site Number 840582, Indianapolis, Indiana
  - Investigational Site Number 840694, Michigan City, Indiana
  - Investigational Site Number 840052, Muncie, Indiana
  - Investigational Site Number 840786, New Albany, Indiana
  - Investigational Site Number 840686, Council Bluffs, Iowa
  - Investigational Site Number 840175, Des Moines, Iowa
  - Investigational Site Number 840466, West Des Moines, Iowa
  - Investigational Site Number 840134, Topeka, Kansas
  - Investigational Site Number 840801, Ashland, Kentucky
  - Investigational Site Number 840754, Benton, Kentucky
  - Investigational Site Number 840342, Covington, Kentucky
  - Investigational Site Number 840713, Elizabethtown, Kentucky
  - Investigational Site Number 840681, Hopkinsville, Kentucky
  - Investigational Site Number 840578, Louisville, Kentucky
  - Investigational Site Number 840478, Owensboro, Kentucky
  - Investigational Site Number 840576, Owensboro, Kentucky
  - Investigational Site Number 840819, Owensboro, Kentucky
  - Investigational Site Number 840645, Paris, Kentucky
  - Investigational Site Number 840741, Versailles, Kentucky
  - Investigational Site Number 840592, Covington, Louisiana
  - Investigational Site Number 840744, Covington, Louisiana
  - Investigational Site Number 840532, Crowley, Louisiana
  - Investigational Site Number 840760, Hammond, Louisiana
  - Investigational Site Number 840463, Lake Charles, Louisiana
  - Investigational Site Number 840675, Marrero, Louisiana
  - Investigational Site Number 840133, Metairie, Louisiana
  - Investigational Site Number 840622, Monroe, Louisiana
  - Investigational Site Number 840147, Natchitoches, Louisiana
  - Investigational Site Number 840609, New Orleans, Louisiana
  - Investigational Site Number 840311, Shreveport, Louisiana
  - Investigational Site Number 840619, Slidell, Louisiana
  - Investigational Site Number 840673, Zachary, Louisiana
  - Investigational Site Number 840387, Bangor, Maine
  - Investigational Site Number 840689, Portland, Maine
  - Investigational Site Number 840534, Baltimore, Maryland
  - Investigational Site Number 840455, Catonsville, Maryland
  - Investigational Site Number 840393, Rockville, Maryland
  - Investigational Site Number 840423, Boston, Massachusetts
  - Investigational Site Number 840117, Alpena, Michigan
  - Investigational Site Number 840289, Detroit, Michigan
  - Investigational Site Number 840053, Essexville, Michigan
  - Investigational Site Number 840150, Flint, Michigan
  - Investigational Site Number 840184, Flint, Michigan
  - Investigational Site Number 840236, Kalamazoo, Michigan
  - Investigational Site Number 840210, Southfield, Michigan
  - Investigational Site Number 840258, Stevensville, Michigan
  - Investigational Site Number 840158, Troy, Michigan
  - Investigational Site Number 840524, Troy, Michigan
  - Investigational Site Number 840033, Olive Branch, Mississippi
  - Investigational Site Number 840302, Bridgeton, Missouri
  - Investigational Site Number 840693, Chesterfield, Missouri
  - Investigational Site Number 840041, Jefferson City, Missouri
  - Investigational Site Number 840711, St Louis, Missouri
  - Investigational Site Number 840753, Billings, Montana
  - Investigational Site Number 840603, Butte, Montana
  - Investigational Site Number 840264, Elkhorn, Nebraska
  - Investigational Site Number 840742, Omaha, Nebraska
  - Investigational Site Number 840294, Henderson, Nevada
  - Investigational Site Number 840087, Henderson, Nevada
  - Investigational Site Number 840664, Las Vegas, Nevada
  - Investigational Site Number 840108, Las Vegas, Nevada
  - Investigational Site Number 840412, Las Vegas, Nevada
  - Investigational Site Number 840656, Las Vegas, Nevada
  - Investigational Site Number 840638, Las Vegas, Nevada
  - Investigational Site Number 840750, Las Vegas, Nevada
  - Investigational Site Number 840815, Las Vegas, Nevada
  - Investigational Site Number 840761, Reno, Nevada
  - Investigational Site Number 840144, Nashua, New Hampshire
  - Investigational Site Number 840799, Edison, New Jersey
  - Investigational Site Number 840167, Linden, New Jersey
  - Investigational Site Number 840060, Neptune City, New Jersey
  - Investigational Site Number 840679, Sicklerville, New Jersey
  - Investigational Site Number 840559, Teaneck, New Jersey
  - Investigational Site Number 840481, Albany, New York
  - Investigational Site Number 840772, Amityville, New York
  - Investigational Site Number 840746, Babylon, New York
  - Investigational Site Number 840355, Brooklyn, New York
  - Investigational Site Number 840136, Brooklyn, New York
  - Investigational Site Number 840734, Forest Hills, New York
  - Investigational Site Number 840659, Great Neck, New York
  - Investigational Site Number 840644, Holbrook, New York
  - Investigational Site Number 840159, Jamaica, New York
  - Investigational Site Number 840148, Lake Success, New York
  - Investigational Site Number 840253, Laurelton, New York
  - Investigational Site Number 840789, Merrick, New York
  - Investigational Site Number 840716, Nesconset, New York
  - Investigational Site Number 840810, New Hyde Park, New York
  - Investigational Site Number 840072, New Hyde Park, New York
  - Investigational Site Number 840674, New Windsor, New York
  - Investigational Site Number 840626, New York, New York
  - Investigational Site Number 840586, New York, New York
  - Investigational Site Number 840044, North Massapequa, New York
  - Investigational Site Number 840587, Smithtown, New York
  - Investigational Site Number 840577, Staten Island, New York
  - Investigational Site Number 840773, Syosset, New York
  - Investigational Site Number 840047, Yonkers, New York
  - Investigational Site Number 840214, Asheville, North Carolina
  - Investigational Site Number 840237, Burlington, North Carolina
  - Investigational Site Number 840714, Burlington, North Carolina
  - Investigational Site Number 840456, Charlotte, North Carolina
  - Investigational Site Number 840312, Concord, North Carolina
  - Investigational Site Number 840763, Greensboro, North Carolina
  - Investigational Site Number 840611, Greensboro, North Carolina
  - Investigational Site Number 840776, Greensboro, North Carolina
  - Investigational Site Number 840361, Greenville, North Carolina
  - Investigational Site Number 840705, High Point, North Carolina
  - Investigational Site Number 840755, Lexington, North Carolina
  - Investigational Site Number 840688, Mooresville, North Carolina
  - Investigational Site Number 840747, Mooresville, North Carolina
  - Investigational Site Number 840296, Morganton, North Carolina
  - Investigational Site Number 840573, New Bern, North Carolina
  - Investigational Site Number 840096, Salisbury, North Carolina
  - Investigational Site Number 840697, Shelby, North Carolina
  - Investigational Site Number 840636, Wilmington, North Carolina
  - Investigational Site Number 840195, Wilson, North Carolina
  - Investigational Site Number 840315, Winston-Salem, North Carolina
  - Investigational Site Number 840545, Fargo, North Dakota
  - Investigational Site Number 840077, Canal Fulton, Ohio
  - Investigational Site Number 840738, Canton, Ohio
  - Investigational Site Number 840064, Cincinnati, Ohio
  - Investigational Site Number 840701, Cincinnati, Ohio
  - Investigational Site Number 840779, Cleveland, Ohio
  - Investigational Site Number 840380, Columbus, Ohio
  - Investigational Site Number 840339, Columbus, Ohio
  - Investigational Site Number 840063, Columbus, Ohio
  - Investigational Site Number 840191, Columbus, Ohio
  - Investigational Site Number 840752, Columbus, Ohio
  - Investigational Site Number 840684, Elyria, Ohio
  - Investigational Site Number 840663, Findlay, Ohio
  - Investigational Site Number 840379, Franklin, Ohio
  - Investigational Site Number 840126, Gallipolis, Ohio
  - Investigational Site Number 840771, Kettering, Ohio
  - Investigational Site Number 840257, Lancaster, Ohio
  - Investigational Site Number 840584, Lyndhurst, Ohio
  - Investigational Site Number 840165, Marion, Ohio
  - Investigational Site Number 840800, Miamisburg, Ohio
  - Investigational Site Number 840560, Tallmadge, Ohio
  - Investigational Site Number 840515, Toledo, Ohio
  - Investigational Site Number 840797, Vandalia, Ohio
  - Investigational Site Number 840192, Wadsworth, Ohio
  - Investigational Site Number 840389, Willoughby Hills, Ohio
  - Investigational Site Number 840751, Wooster, Ohio
  - Investigational Site Number 840262, Edmond, Oklahoma
  - Investigational Site Number 840360, Midwest City, Oklahoma
  - Investigational Site Number 840363, Oklahoma City, Oklahoma
  - Investigational Site Number 840556, Oklahoma City, Oklahoma
  - Investigational Site Number 840103, Bend, Oregon
  - Investigational Site Number 840292, Altoona, Pennsylvania
  - Investigational Site Number 840009, Beaver, Pennsylvania
  - Investigational Site Number 840059, Downingtown, Pennsylvania
  - Investigational Site Number 840181, Fleetwood, Pennsylvania
  - Investigational Site Number 840743, Greensburg, Pennsylvania
  - Investigational Site Number 840479, Huntingdon Valley, Pennsylvania
  - Investigational Site Number 840712, Indiana, Pennsylvania
  - Investigational Site Number 840523, Lansdale, Pennsylvania
  - Investigational Site Number 840766, Levittown, Pennsylvania
  - Investigational Site Number 840032, Penndel, Pennsylvania
  - Investigational Site Number 840067, Philadelphia, Pennsylvania
  - Investigational Site Number 840277, Philadelphia, Pennsylvania
  - Investigational Site Number 840561, Philadelphia, Pennsylvania
  - Investigational Site Number 840174, Philadelphia, Pennsylvania
  - Investigational Site Number 840348, Pittsburgh, Pennsylvania
  - Investigational Site Number 840669, Pottstown, Pennsylvania
  - Investigational Site Number 840748, Sayre, Pennsylvania
  - Investigational Site Number 840187, Smithfield, Pennsylvania
  - Investigational Site Number 840287, Uniontown, Pennsylvania
  - Investigational Site Number 840341, Uniontown, Pennsylvania
  - Investigational Site Number 840378, Providence, Rhode Island
  - Investigational Site Number 840491, Anderson, South Carolina
  - Investigational Site Number 840732, Greenville, South Carolina
  - Investigational Site Number 840043, Greer, South Carolina
  - Investigational Site Number 840109, Murrells Inlet, South Carolina
  - Investigational Site Number 840327, North Myrtle Beach, South Carolina
  - Investigational Site Number 840759, Simpsonville, South Carolina
  - Investigational Site Number 840628, Summerville, South Carolina
  - Investigational Site Number 840717, Bristol, Tennessee
  - Investigational Site Number 840160, Chattanooga, Tennessee
  - Investigational Site Number 840794, Franklin, Tennessee
  - Investigational Site Number 840171, Jackson, Tennessee
  - Investigational Site Number 840550, Jackson, Tennessee
  - Investigational Site Number 840132, Kingsport, Tennessee
  - Investigational Site Number 840140, Knoxville, Tennessee
  - Investigational Site Number 840625, Memphis, Tennessee
  - Investigational Site Number 840299, Nashville, Tennessee
  - Investigational Site Number 840381, New Tazewell, Tennessee
  - Investigational Site Number 840213, Amarillo, Texas
  - Investigational Site Number 840157, Corpus Christi, Texas
  - Investigational Site Number 840011, Dallas, Texas
  - Investigational Site Number 840313, Dallas, Texas
  - Investigational Site Number 840013, Dallas, Texas
  - Investigational Site Number 840034, Dallas, Texas
  - Investigational Site Number 840333, Dallas, Texas
  - Investigational Site Number 840405, Dallas, Texas
  - Investigational Site Number 840330, El Paso, Texas
  - Investigational Site Number 840307, Fort Worth, Texas
  - Investigational Site Number 840182, Houston, Texas
  - Investigational Site Number 840366, Houston, Texas
  - Investigational Site Number 840608, Houston, Texas
  - Investigational Site Number 840323, Houston, Texas
  - Investigational Site Number 840502, Houston, Texas
  - Investigational Site Number 840513, Houston, Texas
  - Investigational Site Number 840377, Houston, Texas
  - Investigational Site Number 840306, Houston, Texas
  - Investigational Site Number 840137, Houston, Texas
  - Investigational Site Number 840521, Houston, Texas
  - Investigational Site Number 840533, Houston, Texas
  - Investigational Site Number 840211, Houston, Texas
  - Investigational Site Number 840260, Humble, Texas
  - Investigational Site Number 840403, Irving, Texas
  - Investigational Site Number 840382, Lampasas, Texas
  - Investigational Site Number 840680, Lubbock, Texas
  - Investigational Site Number 840308, McAllen, Texas
  - Investigational Site Number 840549, Mesquite, Texas
  - Investigational Site Number 840351, Missouri City, Texas
  - Investigational Site Number 840373, Palestine, Texas
  - Investigational Site Number 840365, Pharr, Texas
  - Investigational Site Number 840439, Plano, Texas
  - Investigational Site Number 840707, Port Arthur, Texas
  - Investigational Site Number 840692, Richmond, Texas
  - Investigational Site Number 840431, San Antonio, Texas
  - Investigational Site Number 840074, San Antonio, Texas
  - Investigational Site Number 840691, San Antonio, Texas
  - Investigational Site Number 840176, San Antonio, Texas
  - Investigational Site Number 840135, San Antonio, Texas
  - Investigational Site Number 840018, San Antonio, Texas
  - Investigational Site Number 840434, San Antonio, Texas
  - Investigational Site Number 840390, San Antonio, Texas
  - Investigational Site Number 840207, Schertz, Texas
  - Investigational Site Number 840615, Sealy, Texas
  - Investigational Site Number 840097, Sugar Land, Texas
  - Investigational Site Number 840460, Sugar Land, Texas
  - Investigational Site Number 840514, Sugar Land, Texas
  - Investigational Site Number 840530, Sugar Land, Texas
  - Investigational Site Number 840008, Waco, Texas
  - Investigational Site Number 840593, Waco, Texas
  - Investigational Site Number 840809, Waxahachie, Texas
  - Investigational Site Number 840651, Webster, Texas
  - Investigational Site Number 840392, Clinton, Utah
  - Investigational Site Number 840228, Salt Lake City, Utah
  - Investigational Site Number 840189, St. George, Utah
  - Investigational Site Number 840765, West Jordan, Utah
  - Investigational Site Number 840806, West Jordan, Utah
  - Investigational Site Number 840580, Chatham, Virginia
  - Investigational Site Number 840590, Chesapeake, Virginia
  - Investigational Site Number 840788, Danville, Virginia
  - Investigational Site Number 840706, Danville, Virginia
  - Investigational Site Number 840736, Danville, Virginia
  - Investigational Site Number 840575, Fredericksburg, Virginia
  - Investigational Site Number 840662, Hampton, Virginia
  - Investigational Site Number 840795, Lynchburg, Virginia
  - Investigational Site Number 840605, Martinsville, Virginia
  - Investigational Site Number 840620, Newport News, Virginia
  - Investigational Site Number 840088, Norfolk, Virginia
  - Investigational Site Number 840247, North Chesterfield, Virginia
  - Investigational Site Number 840730, Pennington Gap, Virginia
  - Investigational Site Number 840179, Richmond, Virginia
  - Investigational Site Number 840076, Salem, Virginia
  - Investigational Site Number 840354, Virginia Beach, Virginia
  - Investigational Site Number 840704, Winchester, Virginia
  - Investigational Site Number 840709, Everett, Washington
  - Investigational Site Number 840238, Federal Way, Washington
  - Investigational Site Number 840588, Vancouver, Washington
  - Investigational Site Number 840084, Walla Walla, Washington
  - Investigational Site Number 840658, Charleston, West Virginia
  - Investigational Site Number 840595, Lewisburg, West Virginia
- Canada (20):
  - Investigational Site Number 124002, Barrie
  - Investigational Site Number 124005, Brampton
  - Investigational Site Number 124001, Brampton
  - Investigational Site Number 124030, Burlington
  - Investigational Site Number 124017, Calgary
  - Investigational Site Number 124013, Concord
  - Investigational Site Number 124018, Etobicoke
  - Investigational Site Number 124014, Etobicoke
  - Investigational Site Number 124026, Guelph
  - Investigational Site Number 124008, Hamilton
  - Investigational Site Number 124027, Hamilton
  - Investigational Site Number 124010, London
  - Investigational Site Number 124015, Markham
  - Investigational Site Number 124020, Montreal
  - Investigational Site Number 124016, Newmarket
  - Investigational Site Number 124024, Oakville
  - Investigational Site Number 124029, Saint-Laurent
  - Investigational Site Number 124007, Surrey
  - Investigational Site Number 124003, Toronto
  - Investigational Site Number 124025, Vancouver

REFERENCES:
- [Derived] Anderson J, Meneghini L, Hinnen D, Gill J, Coudert M, Evenou P, Munshi M. Target attainment in insulin-naive patients at high risk for hypoglycemia: Results from ACHIEVE Control. J Diabetes Complications. 2021 Apr;35(4):107831. doi: 10.1016/j.jdiacomp.2020.107831. Epub 2020 Dec 31. PMID 33509703
- [Derived] Oster G, Sullivan SD, Dalal MR, Kazemi MR, Rojeski M, Wysham CH, Sung J, Johnstone B, Cali AM, Wei LJ, Traylor L, Anhalt H, Hull M, Van Vleet J, Meneghini LF. Achieve control: a pragmatic clinical trial of insulin glargine 300 U/mL versus other basal insulins in insulin-naive patients with type 2 diabetes. Postgrad Med. 2016 Nov;128(8):731-739. doi: 10.1080/00325481.2016.1241663. Epub 2016 Oct 24. PMID 27690710

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 427 sites in 2 countries. A total of 4989 participants were screened between 16 June 2015 and 14 July 2017, of which 1684 were screen failures. Screen failures were mainly due to inclusion criteria not met.
Pre-assignment Details: Out of 3305 participants, 1 participant was not randomized, but received treatment; hence not included in any analysis (baseline, efficacy and safety). Assignment in arms was done centrally by interactive response technology (IRT) in 1:1 ratio.
Groups:
- Toujeo: Toujeo® (Insulin glargine, 300 units per millilitre [U/mL]) subcutaneous (SC) injection administered once daily up to Month 12, with or without available participant support program.
Period: Overall Study
Arm/Group | Toujeo | Standard of Care
Started | 1651 | 1653
Treated | 1632 | 1626
Safety Population (Randomized participants who received atleast 1 dose of drug analyzed according to treatment received) | 1637 (4 participants received Standard of Care instead of Toujeo.) | 1621 (9 participants received Toujeo instead of Standard of Care.)
Completed (Completed 12 month on treatment period(time from 1st IMP intake upto last IMP + 1 day)) | 1405 | 1355
Not Completed | 246 | 298
Not completed — Randomized but not treated | 19 | 27
Not completed — Adverse Event | 43 | 42
Not completed — Lack of Efficacy | 4 | 9
Not completed — Participant decision:discontinue insulin | 41 | 43
Not completed — Hypoglycemia | 2 | 1
Not completed — Investigator's decision | 23 | 19
Not completed — Lost to Follow-up | 53 | 61
Not completed — Physician Decision | 6 | 5
Not completed — Sponsor decision | 13 | 25
Not completed — Withdrawal by Subject | 40 | 63
Not completed — Other than specified above | 2 | 3

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants. Participants belonging to more than one race, have been reported under each applicable category.
Groups:
- Toujeo: Toujeo® (Insulin glargine, 300 U/mL) SC injection once daily up to Month 12, with or without available participant support program.
- Total: Total of all reporting groups
Arm/Group | Toujeo | Standard of Care | Total
Number analyzed (Participants) | 1651 | 1653 | 3304
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (10.8) | 59.1 (11.0) | 59.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 747 | 731 | 1478
  Male | 904 | 922 | 1826
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 286 | 305 | 591
  Not Hispanic or Latino | 1365 | 1348 | 2713
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White | 1283 | 1299 | 2582
  Black | 262 | 238 | 500
  Asian/Oriental | 83 | 95 | 178
  American Indian or Alaska Native | 15 | 12 | 27
  Native Hawaiian or other Pacific Islander | 6 | 4 | 10
  Other | 12 | 14 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 82 | 85 | 167
  United States | 1569 | 1568 | 3137
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Here, number analyzed = participants with available data for specified measure.
  kg/m^2
    number analyzed (Participants) | 1649 | 1652 | 3301
    (all) | 33.85 (7.14) | 33.70 (7.29) | 33.77 (7.22)
Duration of Type 2 Diabetes Mellitus [Mean (Standard Deviation); unit: years] | 11.43 (7.43) | 11.16 (7.31) | 11.30 (7.37)
Baseline glycated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] | 9.1 (0.8) | 9.2 (0.8) | 9.2 (0.8)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Individualized Glycated Hemoglobin Target Attainment Per Healthcare Effectiveness Data and Information Set (HEDIS) Criteria Without Documented Symptomatic(Blood Glucose <=70 mg/dL [<=3.9 mmol/L]) and/or Severe Hypoglycemia
Description: HEDIS criteria: Individualized HbA1c target <8% if age >= 65 years or presence of medical comorbidities, or otherwise <7%. Severe hypoglycaemia was an event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Documented symptomatic hypoglycaemia was an event during which typical symptoms of hypoglycaemia were accompanied by a measured plasma glucose concentration of <=70 milligrams per deciliter (mg/dL) (<=3.9 millimoles per litre [mmol/L]). Analysis was performed using all post-baseline data available on the 6 month randomized period (defined as time from randomization up to Day 180 or discontinuation date, whichever comes earlier).
Time Frame: Baseline to Month 6
Population: Analysis was performed on Intent-to-Treat (ITT) population which comprised of all randomized participants, irrespective of the treatment actually received, and analyzed according to the treatment group allocated by randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Toujeo | Standard of Care
Number analyzed (Participants) | 1651 | 1653
percentage of participants | 31.3 | 27.9
Statistical Analysis 1: Comparison: Toujeo vs Standard of Care; A logistic regression model was used with treatment arm as a fixed effect and adjusted for: randomization strata of HbA1c target (<8%,<7%), sulfonylurea (SU) use (yes/no), glucagon like peptide1-receptor agonists (GLP-1 RA) use (yes/no) and baseline HbA1c (as continuous); Test type: Superiority; p = 0.0308, Regression, Logistic — Threshold for significance at 0.046 level; Odds Ratio (OR) = 1.19, 95.4% CI 2-sided [1.01 to 1.39]

2. Secondary Outcome: Change From Baseline in HbA1c at Month 6 and Month 12
Description: Change in HbA1c was calculated by subtracting baseline value from Month 6 and Month 12 values. Adjusted Least Squares (LS) means and Standard Errors (SE) were obtained using Mixed Effect Model with Repeated Measures (MMRM ) with fixed categorical effects of treatment arm, visit, treatment arm-by-visit interaction, randomization strata of HbA1c target (<8% / <7%), SU use (yes/no), GLP-1 RA use (yes/no), as well as baseline HbA1c (as continuous) and baseline HbA1c-by-visit interaction.
Time Frame: Baseline, Month 6, Month 12
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Toujeo | Standard of Care
Number analyzed (Participants) | 1651 | 1653
percentage of HbA1c
  Month 6 | -1.40 (0.030) | -1.36 (0.030)
  Month 12 | -1.29 (0.034) | -1.24 (0.034)

3. Secondary Outcome: Treatment Persistence Measured by Medication Possession Ratio (MPR)
Description: Treatment persistence was determined based on vendor claims database that would be responsible for managing and administration of the study drugs. Medication use was assessed by MPR and persistence measures based on data collected by the smart card vendor (date of fill or refill and quantity of medication dispensed for 30-day supply). The MPR was assessed based on total number of days of supply divided by the total number of days in 6 or 12 months period.
Time Frame: At Month 6 and Month 12
Population: Analysis was performed on safety population.
Measure: Mean (Standard Deviation); unit: Medication Possession ratio
Arm/Group | Toujeo | Standard of Care
Number analyzed (Participants) | 1637 | 1621
Medication Possession ratio
  Month 6 | 62.06 (26.98) | 63.14 (28.42)
  Month 12 | 58.21 (28.87) | 57.82 (29.97)

4. Secondary Outcome: Percentage of Participants Reaching Individualized HbA1c Target Without Documented Symptomatic <3.0 mmol/L (<54 mg/dL) and/or Severe Hypoglycemia During the 6-Month Randomized Period
Description: HEDIS criteria for Individualized HbA1c target: <8% if age >= 65 years or presence of medical comorbidities, or otherwise <7%. Severe hypoglycaemia was an event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Documented symptomatic hypoglycaemia was an event during which typical symptoms of hypoglycaemia were accompanied by a measured plasma glucose concentration of <54 mg/dL (3.0 mmol/L).
Time Frame: Baseline to Month 6
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Toujeo | Standard of Care
Number analyzed (Participants) | 1651 | 1653
percentage of participants | 37.3 | 34.3

5. Secondary Outcome: Percentage of Participants Reaching Individualized HbA1c Target Without Documented Symptomatic <=3.9 mmol/L (<= 70 mg/dL) and <3.0 mmol/L (< 54 mg/dL) and/or Severe Hypoglycemia During the 12-Month Randomized Period
Description: HEDIS criteria for Individualized HbA1c target: <8% if age >= 65 years or presence of medical comorbidities, or otherwise <7%. Severe hypoglycaemia was an event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Documented symptomatic hypoglycaemia was an event during which typical symptoms of hypoglycaemia were accompanied by a measured plasma glucose concentration of <=3.9 mmol/L (<=70 mg/dL) and < 3.0 mmol/L (< 54 mg/dL).
Time Frame: Baseline to Month 12
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Toujeo | Standard of Care
Number analyzed (Participants) | 1651 | 1653
percentage of participants
  Month 12: <=70 mg/dL | 26.1 | 23.7
  Month 12: <54 mg/dL | 33.0 | 29.5

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Month 6 and Month 12
Description: Change in FPG was calculated by subtracting baseline value from Month 6 and Month 12 values. Adjusted LS means and SE were obtained using MMRM model with fixed categorical effects of treatment arm, randomization strata of HbA1c target (<8% / <7%), SU use (yes/no), GLP-1 RA use (yes/no), as well as baseline FPG (as continuous) and baseline FPG-by-visit interaction.
Time Frame: Baseline, Month 6, Month 12
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Toujeo | Standard of Care
Number analyzed (Participants) | 1651 | 1653
mg/dL
  Month 6 | -48.9 (1.56) | -50.4 (1.58)
  Month 12 | -48.0 (1.66) | -47.3 (1.69)

7. Secondary Outcome: Change From Baseline in Body Weight at Month 6 and Month 12
Description: Adjusted LS means and SE were obtained using MMRM model with fixed categorical effects of treatment arm, visit, treatment arm-by-visit interaction, randomization strata of HbA1c target (<8% / <7%), SU use (yes/no), GLP-1 RA use (yes/no), as well as baseline weight (as continuous) and baseline weight-by-visit interaction.
Time Frame: Baseline, Month 6, Month 12
Population: Analysis was performed on ITT population.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Toujeo | Standard of Care
Number analyzed (Participants) | 1651 | 1653
kilogram (kg)
  Month 6 | 1.02 (0.109) | 1.14 (0.110)
  Month 12 | 1.51 (0.140) | 1.40 (0.142)

8. Secondary Outcome: Change From Baseline in Basal Insulin Dose at Month 6 and Month 12
Description: Change in basal insulin dose was calculated by subtracting baseline value from Month 6 and Month 12 values.
Time Frame: Baseline, Month 6, Month 12
Population: Analysis was performed on safety population. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: Unit/kg (U/kg)
Arm/Group | Toujeo | Standard of Care
Number analyzed (Participants) | 1637 | 1621
Unit/kg (U/kg)
  Month 6: number analyzed (Participants) | 1494 | 1451
  Month 6 | 0.179 (0.212) | 0.183 (0.218)
  Month 12: number analyzed (Participants) | 1384 | 1338
  Month 12 | 0.222 (0.232) | 0.224 (0.241)

9. Secondary Outcome: Percentage of Responders (Participants and Provider) Who Reported "Excellent" or "Good" Responses to Global Effectiveness Scale (GES) Question at Month 6, and Month 12
Description: Participant and Physician (Provider) reported GES for this diabetes study. The GES assessed impact of treatment on scale ranges as: excellent (complete control of diabetes), good (marked improvement of diabetes), moderate (discernible, but limited improvement in diabetes), poor (no appreciable change in diabetes), or worsening of condition (worsening of diabetes). There was no score expressed by numbers and no change measured over the time of the study. Percentage of participants and providers who reported "excellent" or "good" on the GES at Month 6 and Month 12 are reported here.
Time Frame: At Month 6, Month 12
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of responders
Arm/Group | Toujeo | Standard of Care
Number analyzed (Participants) | 1651 | 1653
percentage of responders
  Percentage of Participants: Month 6 | 67.2 | 65.6
  Percentage of Providers: Month 6 | 62.1 | 57.7
  Percentage of Participants: Month 12 | 64.7 | 64.2
  Percentage of Providers: Month 12 | 58.8 | 56.3

10. Secondary Outcome: Scores of Total Treatment Satisfaction, Hyperglycemia Perception, and Hypoglycemia Perception From Diabetes Treatment Satisfaction Questionnaire Status Version (DTSQs) at Baseline, Month 6, Month 12
Description: DTSQs is a validated questionnaire to assess participant's satisfaction with their diabetes treatment. It consists of 8 items, each answered on a Likert scale of 0 to 6. Responses of 6 questions (Items 1, 4, 5, 6, 7 and 8) were summarized to derive total treatment satisfaction score, such that a higher score was indicative of better satisfaction. Total treatment satisfaction score is the sum of items 1, 4-8 scores and ranged from 0 (no satisfaction) to 36 (improvement in treatment satisfaction). Item 2 and Item 3 scores were used for hyperglycemia perception and hypoglycemia perception respectively, where lower scores indicated better health outcome. Perceived frequency of hyperglycemia score (Item 2) and perceived frequency of hypoglycemia score (Item 3) range from 0 (none of the time) to 6 (most of time), where lower scores indicated more satisfaction/better health outcome.
Time Frame: At Baseline, Month 6, Month 12
Population: Analysis was performed on ITT population. Here, "number analyzed" = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Toujeo | Standard of Care
Number analyzed (Participants) | 1651 | 1653
score on a scale
  Total treatment satisfaction score:Baseline: number analyzed (Participants) | 1626 | 1627
  Total treatment satisfaction score:Baseline | 26.5 (7.0) | 26.4 (7.1)
  Total treatment satisfaction score: Month 6: number analyzed (Participants) | 1442 | 1415
  Total treatment satisfaction score: Month 6 | 31.0 (5.5) | 31.1 (5.3)
  Total treatment satisfaction score: Month 12: number analyzed (Participants) | 1331 | 1291
  Total treatment satisfaction score: Month 12 | 30.9 (6.0) | 30.7 (6.1)
  Perceived frequencyof hyperglycemia score:Baseline: number analyzed (Participants) | 1625 | 1630
  Perceived frequencyof hyperglycemia score:Baseline | 4.3 (1.7) | 4.3 (1.7)
  Perceived frequency of hyperglycemia score:Month 6: number analyzed (Participants) | 1440 | 1404
  Perceived frequency of hyperglycemia score:Month 6 | 2.8 (1.7) | 2.8 (1.7)
  Perceived frequency of hyperglycemia score:Month12: number analyzed (Participants) | 1326 | 1291
  Perceived frequency of hyperglycemia score:Month12 | 2.6 (1.7) | 2.6 (1.7)
  Perceived frequency of hypoglycemia score:Baseline: number analyzed (Participants) | 1626 | 1630
  Perceived frequency of hypoglycemia score:Baseline | 0.9 (1.4) | 0.8 (1.3)
  Perceived frequency of hypoglycemia score: Month 6: number analyzed (Participants) | 1439 | 1403
  Perceived frequency of hypoglycemia score: Month 6 | 0.9 (1.3) | 1.0 (1.4)
  Perceived frequency of hypoglycemia score:Month 12: number analyzed (Participants) | 1326 | 1288
  Perceived frequency of hypoglycemia score:Month 12 | 0.9 (1.3) | 1.0 (1.4)

11. Secondary Outcome: Scores of Total Treatment Satisfaction, Hyperglycemia Perception, and Hypoglycemia Perception From Diabetes Treatment Satisfaction Questionnaire Change Version (DTSQc) at Month 12
Description: DTSQc version evaluates the change in treatment satisfaction at Month 12 as compared to the start of the study . It consists of 8 items, each answered on a Likert scale from -3 to +3. The sum of treatment satisfaction scores (items 1, 4, 5, 6, 7,and 8) ranged from score -18 (deterioration in treatment satisfaction) to +18 (improvement in treatment satisfaction). Perceived frequency of hypoglycemia and perceived frequency of hyperglycemia score ranges from score -3 (fewer problems) to +3 (more problems).
Time Frame: At Month 12
Population: Analysis was performed on ITT population. Here, "number analyzed" = participants with available data for assessment during the 12 month randomized period.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Toujeo | Standard of Care
Number analyzed (Participants) | 1651 | 1653
score on a scale
  Total satisfaction score: number analyzed (Participants) | 1347 | 1312
  Total satisfaction score | 13.81 (0.15) | 13.79 (0.15)
  Perceived frequency of hyperglycemia score: number analyzed (Participants) | 1341 | 1300
  Perceived frequency of hyperglycemia score | 0.14 (0.05) | 0.21 (0.05)
  Perceived frequency of hypoglycemia: number analyzed (Participants) | 1337 | 1299
  Perceived frequency of hypoglycemia | -0.82 (0.05) | -0.82 (0.05)

12. Secondary Outcome: Percentage of Participants With Hospitalizations, Emergency Rooms and Specialty Visits From Baseline to Month 6 and Month 12
Description: Percentage of participants with hospitalizations, emergency room visits, and specialty visits during the 6-month and 12-month randomized period were reported. The 12-month randomized period was defined as the time from randomization up to Day 365 or discontinuation date, whichever comes earlier.
Time Frame: From Baseline to Month 6 and Month 12
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Toujeo | Standard of Care
Number analyzed (Participants) | 1651 | 1653
percentage of participants
  Hospitalizations: Month 6 | 8.1 | 7.5
  Emergency Room Visits: Month 6 | 11.3 | 10.3
  Specialty Visits: Month 6 | 78.3 | 74.0
  Hospitalizations: Month 12 | 9.1 | 8.0
  Emergency Room Visits: Month 12 | 12.7 | 11.1
  Specialty Visits: Month 12 | 80.1 | 75.9

13. Secondary Outcome: Percentage of Participants With at Least One Treatment-Emergent Hypoglycemia Event (Any Time of the Day, Nocturnal) Per Type of Hypoglycaemia During the Month 6 and Month 12 on Treatment Period
Description: Severe hypoglycaemia was an event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Documented symptomatic hypoglycaemia was an event during which typical symptoms of hypoglycaemia were accompanied by a measured plasma glucose concentration of <=70 mg/dL (<=3.9 mmol/L) or <54 mg/dL (3.0 mmol/L).
Time Frame: Up to Month 6 and Month 12
Population: Analysis was performed on safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Toujeo | Standard of Care
Number analyzed (Participants) | 1637 | 1621
percentage of participants
  Any hypoglycemia: Any time: Month 6 | 28.9 | 30.4
  Any hypoglycemia: Nocturnal: Month 6 | 8.9 | 10.0
  Any hypoglycemia: Any time: Month 12 | 39.1 | 41.8
  Any hypoglycemia: Nocturnal: Month 12 | 13.6 | 14.9
  Severe hypoglycemia: Any time: Month 6 | 1.0 | 1.0
  Severe hypoglycemia:Nocturnal: Month 6 | 0.5 | 0.6
  Documented Symptomatic <=70 mg/dL:Any time:Month 6 | 13.9 | 14.9
  Documented Symptomatic <54 mg/dL:Any time:Month 6 | 3.6 | 3.1
  Documented Symptomatic <=70mg/dL:Nocturnal:Month 6 | 4.5 | 5.6
  Documented Symptomatic <54 mg/dL:Nocturnal:Month 6 | 0.8 | 0.8
  Severe hypoglycemia: Any time: Month 12 | 1.2 | 1.9
  Severe hypoglycemia:Nocturnal: Month 12 | 0.5 | 0.7
  Documented Symptomatic<=70 mg/dL:Any time:Month 12 | 19.9 | 20.8
  Documented Symptomatic <54 mg/dL:Any time:Month 12 | 5.6 | 5.6
  Documented Symptomatic<=70mg/dL:Nocturnal:Month 12 | 6.5 | 8.3
  Documented Symptomatic <54mg/dL:Nocturnal:Month 12 | 1.2 | 1.7

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the end of study (12 months) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (time from the first injection of investigational medicinal product (IMP) up to 1 day after the last injection of IMP). Analysis was performed on safety population.
Groups:
- Standard of Care Basal Insulin: Lantus® (Insulin glargine, 100 U/mL) SC injection administered once daily; or Levemir® (insulin detemir) SC injection administered either once or twice daily up to Month 12, with or without available participant support program.
Arm/Group | Toujeo | Standard of Care Basal Insulin
All-Cause Mortality (participants affected / at risk) | 7/1637 | 4/1621
Serious Adverse Events (participants affected / at risk) | 161/1637 | 165/1621
Other Adverse Events (participants affected / at risk) | 0/1637 | 0/1621
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Toujeo (N=1637) | Standard of Care Basal Insulin (N=1621)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy Mediastinal (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute Left Ventricular Failure (Cardiac disorders) | 3 (3) | 2 (2)
Acute Myocardial Infarction (Cardiac disorders) | 8 (8) | 4 (4)
Angina Pectoris (Cardiac disorders) | 6 (7) | 3 (3)
Angina Unstable (Cardiac disorders) | 4 (5) | 4 (4)
Aortic Valve Stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 (1) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 8 (8) | 6 (6)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular Block Complete (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Bundle Branch Block Left (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Acute (Cardiac disorders) | 4 (4) | 3 (3)
Cardiac Failure Congestive (Cardiac disorders) | 6 (6) | 4 (4)
Coronary Artery Disease (Cardiac disorders) | 10 (10) | 9 (9)
Coronary Artery Stenosis (Cardiac disorders) | 2 (2) | 1 (1)
Intracardiac Thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic Cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 3 (3) | 3 (3)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Autoimmune Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 0 (0)
Retinal Haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2)
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large Intestine Polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis Necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Varices Oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (1) | 1 (2)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0)
Gait Disturbance (General disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 10 (10) | 5 (5)
Pelvic Mass (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Sudden Death (General disorders) | 0 (0) | 1 (1)
Systemic Inflammatory Response Syndrome (General disorders) | 1 (1) | 2 (2)
Vascular Stent Stenosis (General disorders) | 0 (0) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1) | 1 (1)
Biliary Dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 3 (3)
Cirrhosis Alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 2 (2)
Sarcoidosis (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Appendicitis Perforated (Infections and infestations) | 0 (0) | 1 (1)
Arthritis Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Breast Abscess (Infections and infestations) | 0 (0) | 1 (1)
Breast Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 7 (7)
Cholecystitis Infective (Infections and infestations) | 0 (0) | 2 (2)
Cystitis (Infections and infestations) | 1 (1) | 1 (1)
Diabetic Foot Infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 1 (1)
Escherichia Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Escherichia Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0)
Infectious Colitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Localised Infection (Infections and infestations) | 0 (0) | 1 (1)
Ludwig Angina (Infections and infestations) | 1 (1) | 0 (0)
Necrotising Fasciitis (Infections and infestations) | 0 (0) | 2 (2)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1)
Osteomyelitis Acute (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis Chronic (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 10 (10) | 14 (14)
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 1 (1) | 0 (0)
Pseudomembranous Colitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 8 (8)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary Tract Infection Staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Animal Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Endotracheal Intubation Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skull Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ureteric Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram Qt Prolonged (Investigations) | 0 (0) | 1 (1)
Electrocardiogram St Segment Elevation (Investigations) | 1 (1) | 0 (0)
Liver Function Test Increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid Overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperglycaemic Hyperosmolar Nonketotic Syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neuropathic Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma Of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Benign Neoplasm Of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign Ovarian Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder Transitional Cell Carcinoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear Cell Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Malignant Neoplasm Of Ampulla Of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases To Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neurilemmoma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oesophageal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian Epithelial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Peripheral T-Cell Lymphoma Unspecified Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Spindle Cell Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous Cell Carcinoma Of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tonsil Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Arachnoiditis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid Arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Atrophy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 6 (6) | 3 (3)
Cervical Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Focal Dyscognitive Seizures (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic Unconsciousness (Nervous system disorders) | 1 (1) | 2 (3)
Ischaemic Stroke (Nervous system disorders) | 2 (2) | 0 (0)
Lacunar Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Lateral Medullary Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic Encephalopathy (Nervous system disorders) | 2 (2) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Nerve Compression (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (3) | 2 (2)
Transient Ischaemic Attack (Nervous system disorders) | 3 (3) | 3 (3)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Device Loosening (Product Issues) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 3 (3)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 8 (8) | 9 (10)
Calculus Bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Diabetic Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 4 (4)
Renal Failure (Renal and urinary disorders) | 3 (3) | 0 (0)
Renal Impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric Obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary Bladder Polyp (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic Foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Necrobiosis Lipoidica Diabeticorum (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Stasis Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pregnancy Of Partner (Social circumstances) | 0 (0) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Brachiocephalic Artery Stenosis (Vascular disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 2 (3) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 (0) | 4 (4)
Peripheral Artery Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Artery Occlusion (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT02451137/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT02451137/SAP_001.pdf